CLINICAL TRIAL: NCT02245139
Title: Surveillance Study of Acute Gastroenteritis Etiologies in Hospitalized Children
Brief Title: Surveillance Study of Acute Gastroenteritis in Hospitalized Children
Acronym: SAGE
Status: Completed | Type: Observational
Sponsor: Shaikh Ragheb Harb Hospital (Other)
Responsible Party: Principal Investigator, HADI FAKIH, MD, MD, Shaikh Ragheb Harb Hospital
Other Study IDs: SRHH12014
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Acute Gastroenteritis; Diarrhea; Dehydration
Keywords: diarrhea; vomiting; fever; abdominal pain; oliguria
MeSH Terms: conditions — Diarrhea; Dehydration; Vomiting; Fever; Abdominal Pain; Oliguria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute gastroenteritis is a common cause of hospital admission and health office visits and have a huge burden on the economy of developing countries. The investigators proposed this observational prospective study during summer period in a community and tertiary care hospital in a rural area of Lebanon to investigate the etiologies and age distribution of admitted cases to general pediatric floor from the age of 1 month up to the age of 14 years.

ELIGIBILITY:
Inclusion Criteria:

* acute gastroenteritis

Exclusion Criteria:

* immunodeficiency
* malnutrition

Ages: 1 Month to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: male and female patient from 1 month to 13 YO admitted to pediatric floor with acute gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
etiologies | 1 year
  to determine the microbial causes of acute gastroenteritis